CLINICAL TRIAL: NCT04733534
Title: SEN-SURVIVORS: An Open-Label Intervention Trial to Reduce Senescence and Improve Frailty in Adult Survivors of Childhood Cancer
Brief Title: An Open-Label Intervention Trial to Reduce Senescence and Improve Frailty in Adult Survivors of Childhood Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SENSURV; U01CA246510 (NIH)
Record Dates: First submitted 2020-12-09; First posted 2021-02-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Frailty; Childhood Cancer
MeSH Terms: conditions — Frailty; Neoplasms | interventions — Dasatinib; Quercetin; peflavit; Flavonoids; fisetin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dasatinib plus Quercetin (Active Comparator): Day 0 (30 per arm, randomization stratified by sex and age)
  At the visit on day 7, blood CD3+ T lymphocyte p16^INK4A mRNA and other markers of inflammation and senescence will be accessed to verify that senescent cells have been cleared by the intervention.
  Post-treatment follow-up will occur on days 60 for (primary endpoints) and day 150 for secondary evaluation. Day 150 will assess the permanence of change after completion of the trial.
  Interventions: Drug: Dasatinib plus Quercetin
- Fisetin (Active Comparator): Day 0 (30 per arm, randomization stratified by sex and age)
  At the visit on day 7, blood CD3+ T lymphocyte p16INK4A mRNA and other markers of inflammation and senescence will be accessed to verify that senescent cells have been cleared by the intervention.
  Post-treatment follow-up will occur on days 60 for (primary endpoints) and day 150 for secondary evaluation. Day 150 to will assess the permanence of change after completion of the trial.
  Interventions: Drug: Fisetin

INTERVENTIONS:
Drug: Dasatinib plus Quercetin — Dasatinib (100 mg/day) plus Quercetin (500 mg twice daily) on days 1, 2, 3, 30, 31, 32 taken orally under observation of the study nurse.
  Other Names: Sprycel; Pentahydroxyflavone; Bioflavonoid,
  Arms: Dasatinib plus Quercetin
Drug: Fisetin — Fisetin (20mg/kg/day) on days 1, 2, 30 and 31 taken orally under observation of the study nurse. Fisetin will be dispensed based on weight of 20 mg/kg/day on the four separate days.
  Arms: Fisetin

SUMMARY:
This is a first-in survivor pilot study with the goal of establishing preliminary evidence of efficacy, safety, and tolerability of two senolytic regimens to reduce markers of cellular senescence (primary outcome: p16^INK4a) and improve frailty (primary outcome: walking speed) in adult survivors of childhood cancer. If successful, this pilot would provide the preliminary evidence needed for a phase 2, randomized, placebo-controlled trial to establish efficacy.

Primary Objective

* The primary aim of this proposal is to test the efficacy of two, short duration senolytic regimens: 1) combination of Dasatinib plus Quercetin and 2) Fisetin alone, to improve walking speed and decrease senescent cell abundance in blood (p16^INKA):
* Primary endpoints of this trial will be change in walking speed and senescent cell abundance in blood (p16^INK4A) determined at baseline and again at 60 days, within an individual arm. Extended follow up at 150 days will assess the permanence of change after completion of the trial. Secondary endpoints of this trial will be effect of intervention on additional measures of frailty (beyond walking speed; Fried criteria) and on other cell senescence markers, markers of inflammation, insulin resistance, bone resorption, and cognitive function.

Secondary Objectives

The secondary aim is to test the safety and tolerability of two different senolytic therapies.

Exploratory Objectives

* To compare the efficacy of the two senolytic regimens in improving walking speed and decreasing senescent cell abundance
* To evaluate the longitudinal pattern in measures of frailty.

DETAILED DESCRIPTION:
Eligible subjects who meet inclusion criteria will be randomized, stratified on sex, 1:1 and age ( ≥40 vs < 40) to receive Dasatinib (100 mg/day) plus Quercetin (500 mg twice daily) on days 1, 2, 3, 30, 31, and 32 taken orally or Fisetin (20 mg/kg/day) alone on days 1, 2, 30 and 31 taken orally. At the visit on day 7, we will assess blood CD3+ T lymphocyte p16^INK4A mRNA and other markers of inflammation and senescence to verify that senescent cells have been cleared by the intervention. Post-treatment follow-up will occur on day 60 (primary endpoints) and day 150 to assess the permanence of change after completion of the trial. Treatment adherence will be confirmed by the study coordinator who will administer the Dasatinib + Quercetin in clinic on days 1, 2, 3, 30, 31, and 32 or Fisetin alone on days 1, 2, 30 and 31.

ELIGIBILITY:
Inclusion Criteria:

* Participant in SJLIFE and > 5 years from diagnosis.
* ≥18 years of age.
* Frail (2 of 4 objectively measured Fried criteria adapted,(excluding self-reported fatigue as a criteria), including abnormal walking speed; muscle strength; activity level; and muscle mass). See Section 5 for details.
* CD3+ T lymphocytes: p16INK4A detected at <34 cycles by RT PCR.
* Agrees to use contraception as Dasatinib is teratogenic.
* Female participant has a negative pregnancy test.
* QTc <450 milliseconds in electrocardiogram.
* Able to take oral medications.

Exclusion Criteria:

* Currently has HIV, Hepatitis B/C, invasive fungal infection
* Anemia or as per clinical judgement.
* Hypersensitivity to study drugs
* New/active malignancy/taking chemotherapy and/or radiation except non-melanoma skin cancers
* Currently taking medications that inhibit or induce CYP3A4 or that are sensitive to substrates or substrates with a narrow therapeutic range for CYP2C8, CYP2C9, or CYP2D6.
* Taking anticoagulants or antimicrobial agents
* Currently taking Quercetin or Fisetin
* Pregnant or nursing at time of enrollment/during the study
* Impaired cognition or motor performance due to congenital defects
* Currently participating in another research intervention to aid walking speed or other measures of frailty including muscle strength; low activity; muscle mass or exhaustion/fatigue
* Participant is a Non-English Speaker
* Uncontrolled pleural/pericardial effusion or ascites
* Subjects on anticoagulant or antiplatelet agents (Warfarin, Clopidogrel [Plavix]; Dipyridamole + Aspirin [Aggrenox]; Ticagrelor [Brilintal]; Prasugrel [Effient]; Ticlopidine [Ticlid]; or other) who are unable or unwilling to reduce or hold therapy prior to and during the 2-3 day drug dosing. Subjects may continue their previous regimen after drug dosing is complete.
* Cognitive impairment defined by IQ <80
* Diagnosis of a psychotic disorder
* Laboratory tests as indicated or as per clinical judgement
* Severe hepatic dysfunction with ALT/AST > 3 times upper limit of normal.
* Total bilirubin > 2 times upper limit of normal.
* eGFR <25 ml/min/1.73m2 or as per clinical judgement.
* Hemoglobin < 7 g/dl; white blood cell count ≤2,000/mm3 (≤2.0 x 109/L) or ≥20,000/mm3 (≥20 x 109/L); platelet count ≤40,000/μL (≤40 x 109/L); absolute neutrophil count ≤1 x 109/L; lymphocyte count <0.3 x 109/L at screening as a marker of poor nutrition
* Fasting glucose >300.
* Participant is unable to ambulate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in walking speed | Baseline
  Walking speed will be measured by having the participant walk 4 meters as fast as he/she can walk. This test will be measured in meters per second.
Change in Walking Speed | Day 30
  Walking speed will be measured by having the participant walk 4 meters as fast as he/she can walk. This test will be measured in meters per second.
Change in Walking Speed | Day 60
  Walking speed will be measured by having the participant walk 4 meters as fast as he/she can walk. This test will be measured in meters per second.
Change in Walking Speed | Day 150
  Walking speed will be measured by having the participant walk 4 meters as fast as he/she can walk. This test will be measured in meters per second.
Senescent cell abundance in blood (p16INK4A) | Baseline
  Following a 12 hour overnight fast, 10 ml blood will be collected in EDTA tubes, processed at St. Jude and shipped to the Kirkland lab for evaluation of CD3+ peripheral blood T lymphocytes (PTBL) p16INK4A mRNA, a biomarker of senescence and chronological aging. CD3+ PTBL will be isolated from whole blood using Whole Blood CD3 Human Microbeads (Miltenyi Biotec, Cat# 130-090-874) by MACS sorting [79]. CD3+ cells will be lysed, mRNA isolated, and p16INK4A expression assayed by RT-PCR using a Taq-man primer-probe system.
Senescent cell abundance in blood (p16INK4A) | Day 7
  Following a 12 hour overnight fast, 10 ml blood will be collected in EDTA tubes, processed at St. Jude and shipped to the Kirkland lab for evaluation of CD3+ peripheral blood T lymphocytes (PTBL) p16INK4A mRNA, a biomarker of senescence and chronological aging. CD3+ PTBL will be isolated from whole blood using Whole Blood CD3 Human Microbeads (Miltenyi Biotec, Cat# 130-090-874) by MACS sorting [79]. CD3+ cells will be lysed, mRNA isolated, and p16INK4A expression assayed by RT-PCR using a Taq-man primer-probe system.
Senescent cell abundance in blood (p16INK4A) | Day 30
  Following a 12 hour overnight fast, 10 ml blood will be collected in EDTA tubes, processed at St. Jude and shipped to the Kirkland lab for evaluation of CD3+ peripheral blood T lymphocytes (PTBL) p16INK4A mRNA, a biomarker of senescence and chronological aging. CD3+ PTBL will be isolated from whole blood using Whole Blood CD3 Human Microbeads (Miltenyi Biotec, Cat# 130-090-874) by MACS sorting [79]. CD3+ cells will be lysed, mRNA isolated, and p16INK4A expression assayed by RT-PCR using a Taq-man primer-probe system
Senescent cell abundance in blood (p16INK4A) | Day 60
  Following a 12 hour overnight fast, 10 ml blood will be collected in EDTA tubes, processed at St. Jude and shipped to the Kirkland lab for evaluation of CD3+ peripheral blood T lymphocytes (PTBL) p16INK4A mRNA, a biomarker of senescence and chronological aging. CD3+ PTBL will be isolated from whole blood using Whole Blood CD3 Human Microbeads (Miltenyi Biotec, Cat# 130-090-874) by MACS sorting [79]. CD3+ cells will be lysed, mRNA isolated, and p16INK4A expression assayed by RT-PCR using a Taq-man primer-probe system.
Senescent cell abundance in blood (p16INK4A) | Day 150
  Following a 12 hour overnight fast, 10 ml blood will be collected in EDTA tubes, processed at St. Jude and shipped to the Kirkland lab for evaluation of CD3+ peripheral blood T lymphocytes (PTBL) p16INK4A mRNA, a biomarker of senescence and chronological aging. CD3+ PTBL will be isolated from whole blood using Whole Blood CD3 Human Microbeads (Miltenyi Biotec, Cat# 130-090-874) by MACS sorting [79]. CD3+ cells will be lysed, mRNA isolated, and p16INK4A expression assayed by RT-PCR using a Taq-man primer-probe system.

SECONDARY OUTCOMES:
Safety of two different senolytic therapies as assessed by treatment-related adverse events using CTCAE v5.0 | 150 days
  To test the safety of the combination of Dasatinib plus Quercetin or Fisetin alone
Tolerability of two different senolytic therapies as assessed by treatment-related adverse events using CTCAE v5.0 | 150 days
  To test the tolerability of the combination of Dasatinib plus Quercetin or Fisetin alone

CONTACTS AND LOCATIONS:
Overall Officials: Gregory T. Armstrong, MD, MSCE, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols